CLINICAL TRIAL: NCT02055963
Title: Minocycline for Reduction of Symptom Burden After Surgery in Patients With Head and Neck Malignancy: A Randomized Study
Brief Title: Minocycline for Postsurgical Symptom Reduction in Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to the protocol lack of progress in improving accrual rate
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013-0510; R01CA026582 (NIH); NCI-2014-01979 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Head And Neck Cancer
Keywords: Head And Neck Cancer; Postsurgical symptom reduction; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Sugar pill; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms; cyclopia sequence | interventions — Minocycline; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Participants take study medication twice daily, starting 2 days prior to surgery, and continue for 3 weeks postsurgery. The final day of study medication will be the 21st day after surgery.
  Minocycline100 mg given orally every 12 hours on Day -2, (i.e., 2 days prior to surgery) and continuing for 3 weeks postsurgery.
  Questionnaire completion 2 days before surgery, on day of surgery, 1 and 3 days after surgery, then twice a week until follow up visit on day 21.
  Interventions: Drug: Minocycline; Behavioral: Questionnaires
- Placebo (Placebo Comparator): Participants take study medication twice daily, starting 2 days prior to surgery, and continue for 3 weeks postsurgery. The final day of study medication will be the 21st day after surgery.
  Placebo 100 mg given orally every 12 hours on Day -2, (i.e., 2 days prior to surgery).
  Questionnaire completion 2 days before surgery, on day of surgery, 1 and 3 days after surgery, then twice a week until follow up visit on day 21.
  Interventions: Drug: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Minocycline — 100 mg given orally every 12 hours on Day -2, (i.e., 2 days prior to surgery) and continuing for 3 weeks postsurgery.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Drug: Placebo — Placebo 100 mg given orally every 12 hours on Day -2, (i.e., 2 days prior to surgery) and continuing for 3 weeks postsurgery.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Questionnaires — Questionnaire completion 2 days before surgery, on day of surgery, 1 and 3 days after surgery, then twice a week until follow up visit on day 21.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if Minocin® (minocycline) can reduce certain side effects of surgery in patients with head and neck cancer (such as pain, fatigue, and disturbed sleep). In this study, minocycline will be compared to a placebo.

A placebo is not a drug. It looks like the study drug, but it is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being in any group.

* If you are in Group 1, you will receive minocycline.
* If you are in Group 2, you will receive a placebo.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take minocycline/placebo 2 times every day (about 12 hours apart). This will be from 1-2 days before surgery until 3 weeks after surgery.

Most of the time, you will take the minocycline/placebo by mouth or through your feeding tube. If you are unable to take it by mouth or through your feeding tube, you will receive it by vein every 12 hours.

You should take the study drug/placebo with a full glass (8 ounces) of water. You may take it with or without food, but if it causes an upset stomach, you should take it with food.

You should not lie down for at least 30 minutes after taking the study drug/placebo to reduce the risk of side effects.

You will also be given standard drugs to help decrease the risk of side effects from the surgery. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

After you agree to participate in the study, on the day of surgery, 1 and 3 days after surgery, and then about 2 times a week until the end of the study, you will complete a questionnaire about any side effects you are experiencing. This should take about 5 minutes to complete. When you are at home, you will complete this questionnaire over the phone through a computerized system. You will answer the questions using your telephone keypad.

After you agree to participate in the study, and at 1 and 3 days after surgery, you will complete 2 questionnaires about your quality of life. This should take about 10 minutes to complete.

After you agree to participate in the study, soon after your surgery, and 1 week after surgery or when you are discharged from the hospital, saliva will be collected and used to test for markers of inflammation. If possible, blood (about 2 teaspoons) also will be drawn to test for markers of inflammation. This will be during a regular blood draw and you would not need to have an extra needle stick.

Length of Study:

You will take the study drug/placebo for 3 weeks after surgery. You will no longer be able to take the study drug/placebo if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visit.

Follow up Visit:

At about 3 weeks after your surgery, you will return to the clinic. The following tests and procedures will be performed:

* Saliva will be collected and used to test for markers of inflammation.
* You will complete 3 questionnaires about your quality of life and any side effects you are feeling. This should take about 20 minutes to complete.
* If possible, blood (about 2 teaspoons) also will be drawn to test for markers of inflammation. This will be during a regular blood draw and you would not need to have an extra needle stick.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Using minocycline to try to reduce the side effects of surgery in patients with head and neck cancer is investigational.

Up to 130 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and neck cancer who are undergoing either flap or nonflap surgery (limited to parotidectomy, hard palate maxillectomy and glossectomy, mandibulectomy, and any procedure with neck dissection) at MD Anderson Cancer Center.
2. Patients > 18 years old.
3. Patients who have not undergone surgery in the past 6 months. Patients may have had neoadjuvant chemotherapy prior to surgery.
4. Patients must have normal renal function test and no prior renal disease. The screening cut off for serum creatinine is < 1.5mg/dL.
5. Patients must have normal hepatic function test and no prior liver disease: (1) The screening results for alanine aminotransferase (ALT) must be < 2 times the upper limit of normal. (2) The screening results for aspartate aminotransferase (AST), if available, must be < 2 times the upper limit of normal.
6. Patients who speak English or Spanish (due to the novel research and its complexity, we are only accruing English-speaking or Spanish-speaking patients to the protocol).
7. Patients must be willing and able to review, understand, and provide written consent.
8. Patients must be willing to discontinue taking dong quai and/or St. John's wort.

Exclusion Criteria:

1. Patients who are taking medications (including minocycline) or have conditions that potentially preclude use of the study medication or intervention as determined by the treating physician.
2. Patients who are enrolled in another symptom management trial or receiving active treatment under another clinical trial.
3. Patients with a history of clinically significant cutaneous drug reaction, hypersensitivity reaction, anaphylaxis or any other serious adverse reaction to any of the anesthetics or analgesics medications used in the study.
4. Patients with hypersensitivity to any tetracycline.
5. Patients on vitamin K antagonist (i.e., warfarin).
6. Patients taking any tetracycline within the last 15 days.
7. Patients who have been on opioid therapy for the last 4 weeks or more.
8. Patients with bile duct obstruction.
9. Patients who are pregnant.
10. Patients with INR > 1.5.
11. Patients with autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants enrolled at MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Customized [Count of Participants; unit: Participants]
  20 to 29 years | 0 | 1 | 1
  30 to 39 years | 0 | 1 | 1
  40 to 49 years | 2 | 2 | 4
  50 to 59 years | 4 | 2 | 6
  60 to 69 years | 4 | 7 | 11
  70 to 79 years | 4 | 2 | 6
  80 to 89 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 2 | 0 | 2
  White Non-Hispanic | 9 | 15 | 24
  Hispanic | 0 | 1 | 1
  Asian | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Minocycline for Reducing Patient-Reported Symptoms
Description: Primary outcome variable is area under the curve (AUC) using the average of the 3 most severe symptoms (pain, fatigue, and disturbed sleep) beginning 2 days prior to surgery and ending 21 days postsurgery. AUC calculated using trapezoidal approximation. The base of a trapezoid corresponds to the number of days between assessments while the heights correspond to 2 adjoining symptom responses. The number of trapezoids depends on the number of symptom assessments. The sum of the area for all the trapezoids represents the AUC of a particular patient. Data were collected to create the curve (-2, 0, 1, 3, 5, 7, 10, 14, 17, and 21 days post-dose)
Time Frame: -2 to 21 days post-dose
Population: 4 participants were not included in the primary efficacy analysis due to 3 dropped out before 1 week (1 in the Minocycline Arm and 2 in the Placebo Arm) and 1 participants in the Minocycline Arm the MD Anderson Symptom Inventory (MDASI) was not evaluated.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 12 | 14
mcg*hr/mL | 66.4 (32.4) | 67.5 (38.2)
Statistical Analysis 1: Comparison: Minocycline vs Placebo; Test type: Other; p = 0.98, Wilcoxon Rank Sum Test

2. Secondary Outcome: Number of Participants Time-to-Symptom-Recovery
Description: Time-to-symptom-recovery defined to be the time it takes for symptom severity (average of pain, fatigue and disturbed sleep) to return to preoperative levels for 2 consecutive assessments. Repeated measures ANOVA performed with group (minocycline vs. placebo), time (presurgery, postsurgery, discharge, follow up) and group-by-time interaction as factors and proinflammatory cytokine level as a dependent variable. Data measured at Day -2, Day 0, Day 1, Day 3, Day 5, Day 7, Day 10, Day 14, Day 17, Day 20. Cox proportional hazards models were used to explore predictors of time-to-symptom-recovery.
Time Frame: Day -2, Day 0, Day 1, Day 3, Day 5, Day 7, Day 10, Day 14, Day 17, Day 20
Measure: Count of Participants; unit: Participants
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 14 | 16
Participants
  Day -2 | 12 | 14
  Day 0 | 6 | 13
  Day 1 | 11 | 14
  Day 3 | 10 | 13
  Day 5 | 9 | 14
  Day 7 | 10 | 12
  Day 10 | 11 | 12
  Day 14 | 12 | 14
  Day 17 | 11 | 13
  Day 20 | 12 | 14

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study drug medication, up to week 6 ± 1 week post-surgery (in clinic or by phone)
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/16
Other Adverse Events (participants affected / at risk) | 4/14 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=14) | Placebo (N=16)
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=14) | Placebo (N=16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hives (Skin and subcutaneous tissue disorders) | 1 | 0
Itchy (Skin and subcutaneous tissue disorders) | 1 | 0
Lack of appetite (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination due to the protocol lack of progress in improving accrual rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02055963/Prot_SAP_000.pdf